CLINICAL TRIAL: NCT03853109
Title: A Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 404, a Programmed Death-1 (PD-1) Antibody, in Patients With Advanced Solid Tumors
Brief Title: AMG 404 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180143; 2018-004268-80 (EudraCT Number)
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Cohort 1
  Interventions: Drug: AMG 404
- Cohort 2 (Experimental): Cohort 2
  Interventions: Drug: AMG 404
- Cohort 3 (Experimental): Cohort 3
  Interventions: Drug: AMG 404
- Cohort 4 (Experimental): Cohort 4
  Interventions: Drug: AMG 404
- Cohort 6 (Experimental): Cohort 6
  Interventions: Drug: AMG 404
- Cohort 7 (Experimental): Cohort 7
  Interventions: Drug: AMG 404
- Cohort 8 (Experimental): Cohort 8
  Interventions: Drug: AMG 404
- Cohort 9 (Experimental): Cohort 9
  Interventions: Drug: AMG 404

INTERVENTIONS:
Drug: AMG 404 — AMG 404 will be examined for safety, tolerability, PK, and PD of AMG 404 in subjects with advanced solid tumors.

SUMMARY:
To evaluate the safety and tolerability of AMG 404, a monoclonal antibody that binds to PD-1 and inhibits its engagement with ligands, in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study specific activities/procedures.
* Age greater than or equal to 18 years old at the time of signing informed consent.
* Life expectancy of greater than 3 months, in the opinion of the investigator
* Subject must have histologically or cytologically confirmed metastatic or locally advanced solid tumors not amenable to curative treatment with surgery or radiation.
* Cohort 7: participant must have one of the following tumor types: melanoma, small cell lung cancer, NSCLC (PD-L1 positive), head and neck squamous cell cancer (PD-L1 positive), urothelial (PD-L1 positive), gastric or GEJ adenocarcinoma (PD-L1 positive), esophageal (squamous, PD-L1 positive), cervical (PD-L1 positive), hepatocellular carcinoma, merkel cell carcinoma, squamous cell carcinoma of the skin, renal cell carcinoma (clear cell) subtypes of sarcoma (undifferentiated pleiomorphic / malignant fibrous histiocytoma, poorly differentiated and/or dedifferentiated liposarcoma, alveolar soft tissue sarcoma, angiosarcoma), thymic carcinoma, nasopharyngeal carcinoma (EBV positive), mesothelioma
* Cohort 8: participant must be MSI-H or MMR-deficient
* Cohort 9: participant must have NSCLC, PD-L1 positive, TPS ≥ 50%; not have EGFR or ALK or ROS1 genomic tumor aberrations and may not have received prior systemic treatment for the advanced disease (prior neoadjuvant, adjuvant, or concurrent chemoradiation is allowed).
* At least 1 measurable as defined by modified RECIST 1.1 which has not undergone biopsy within 3 months of the screening scan. This lesion cannot be biopsied at any time during the study. Note: if there is only one lesion available for biopsy and radiographic assessment, it may be permitted to be biopsied after discussion with sponsor.
* Subjects with treated brain metastases are eligible provided they meet the following criteria: Definitive therapy was completed at least 2 weeks prior to enrollment. No evidence of radiographic CNS progression or CNS disease following definitive therapy and by the time of study screening. Patients manifesting progression in lesions previously treated with stereotactic radiosurgery may still be eligible if pseudoprogression can be demonstrated by appropriate means and after discussion with the medical monitor.
* Any CNS disease is asymptomatic, any neurologic symptoms due to CNS disease have returned to baseline or are deemed irreversible, the patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the patient is off or on stable doses of anti-epileptic drugs for malignant CNS disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of less than or equal to 2.
* Hematologic function, as follows without growth factor support within 2 weeks prior to study day 1: Absolute neutrophil count (ANC) greater than or equal to 1.0 x 10E9/L; Platelet count greater than or equal to 75 x 10E9/L; Hemoglobin greater than or equal to 9 g/dL (90 g/L).
* Adequate renal laboratory assessments, as follows: Estimated glomerular filtration rate based on MDRD (Modification of Diet in Renal Disease) calculation . 60 ml/min/1.73 m^2 for Cohorts 1, 2, and 4 Estimated glomerular filtration rate based on MDRD (Modification of Diet in Renal Disease) calculation >= 45 ml/min/1.73 m^2 for Cohorts 3, 6, 7, 8 and 9.
* Hepatic function, as follows: Total bilirubin less than or equal to 1.5 x ULN or less than or equal to 3 x ULN for subjects with liver metastasis; AST less than or equal to 3 x ULN or less than or equal to' 5 x ULN for subjects with liver metastasis; ALT less than or equal to 3 x ULN or less than or equal to 5 x ULN for subjects with liver metastasis; Alkaline phosphatase less than or equal to 2.5 x ULN or less than or equal to 5 x ULN for subjects with liver metastasis (Note: elevated alkaline phosphatase is acceptable if it is due to non-hepatic associated pathology [eg, bone disease]).
* Subjects enrolled to Cohorts 7-9 must submit tumor tissue sample. Fresh tumor biopsies may be performed if subject has a readily accessible tumor lesion and who consent to the biopsies. If fresh biopsies cannot be obtained, archival tumor samples are acceptable. Prior to enrollment it is required to determine that there is enough tumor tissue available to be sent to the central laboratory: Cohorts 7 and 9: Archival tissue collected up to 12 months prior to screening date is permitted. Biopsies collected between 12-18 months prior to screening are allowed upon discussion with the medical monitor. Subjects with EBV associated nasopharyngeal carcinoma may submit biopsy with EBV test results from within 36 months prior to screening; Cohort 8: Archival tissue with MSI-high/dMMR test results collected up to 36 months prior to screening is permitted.

Exclusion Criteria:

* Disease Related. Primary brain tumor, untreated or symptomatic brain metastases and leptomeningeal disease (exception: benign asymptomatic tumors are permitted).
* Other Medical Conditions. History of other malignancy within the past 2 years, with the following exception[s]: Malignancy treated with curative intent and with no known active disease present for greater than or equal to 2 years before enrollment and felt to be at low risk for recurrence by the treating physician. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease. Adequately treated cervical carcinoma in situ without evidence of disease. Adequately treated breast ductal carcinoma in situ without evidence of disease. Prostatic intraepithelial neoplasia without evidence of prostate cancer. Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ. Other malignancies which do not require systemic therapy, may be considered upon discussion with the medical monitor.
* History of solid organ transplantation.
* Major surgery within 28 days of study day 1.
* Prior/Concomitant Therapy: Prior treatment with anti-programmed death 1 (PD-1), anti-PD-L1, CTLA-4 or other checkpoint inhibitor drugs
* Anti-tumor therapy (radiotherapy, chemotherapy, antibody therapy, molecular targeted therapy, or investigational agent) within 21 days prior to study day 1. Note: Palliative radiotherapy is permitted.
* Live vaccine therapy within 4 weeks prior to study drug administration.
* Current treatment or within 14 days of day 1 with immunosuppressive corticosteroid defined as greater than 10 mg prednisone daily or equivalent. Corticosteroids with no or minimal systemic effect (such as topical or inhalation) are permitted. Note: Corticosteroids > 10 mg prednisone used for management of contrast allergy for study scans is allowed.
* Prior/Concurrent Clinical Study Experience: Currently receiving treatment in another investigational device or drug study, or less than 21 days prior to study day 1 since ending treatment on another investigational device or drug study(ies).
* Diagnostic Assessments: Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* History of any immune-related colitis. Infectious colitis is allowed if evidence of adequate treatment and clinical recovery exists and at least 3 months interval observed since diagnosis of colitis.
* History of allergic reactions or acute hypersensitivity reaction to antibody therapies.
* Positive/Non-negative test for Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B (eg, hepatitis B antigen [HBsAg] reactive) or Hepatitis C (eg, HCV RNA [qualitative] is detected).
* Subject currently has an active infection requiring systemic therapy.
* Active or history of any autoimmune disease or immunodeficiencies. Subjects with Type I diabetes, vitiligo, psoriasis, hypo- or hyper- thyroid disease not requiring immunosuppressive treatment are permitted.
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association greater than class II), unstable angina, or cardiac arrhythmia requiring antiarrhythmic medication.
* Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1, or are stable and well controlled with minimal, local, or non-invasive intervention AND there is agreement to allow by both the investigator and the Amgen Medical Monitor.
* Other Exclusions: Males and females of reproductive potential who are unwilling to practice highly effective methods of birth control while on study through 6 months (females) and 8 months (males) after receiving the last dose of AMG 404.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (34):
- United States (5):
  - Sarcoma Oncology Research Center LLC, Santa Monica, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- Brazil (5):
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
  - Instituto Coi, Rio de Janeiro
- Tom Baker Cancer Centre, Calgary, Alberta, Canada
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (2):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Universitario La Paz, Madrid
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Turkey (Türkiye) (3):
  - Doktor Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Koc Universitesi Hastanesi, Istanbul
  - Ege Universitesi Ilac Gelistirme ve Farmakokinetik Arastirma Uygulama Merkezi (ARGEFAR), Izmir
- Sarah Cannon Research Institute UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Price T, Lugowska I, Chawla SP, Falchook G, Subbiah V, Monzon JG, Arkenau HT, Hui M, Kuboki Y, Dziadziuszko R, Shibaki R, Hong MH, Tan D, Rocha Lima CM, Wang K, Hindoyan A, Shi W, Wong H, Kistler M, Prenen H. A phase I, open-label, multicentre, first-in-human study to evaluate safety, pharmacokinetics and efficacy of AMG 404, a PD-1 inhibitor, in patients with advanced solid tumours. BMJ Open. 2025 May 2;15(5):e088578. doi: 10.1136/bmjopen-2024-088578. PMID 40316348
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 34 centers in Australia, Belgium, Brazil, Canada, Japan, Poland, Singapore, South Korea, Spain, Taiwan, Turkey, the United Kingdom, and the United States. Participants were recruited between 05 March 2019 and 02 November 2023.
Pre-assignment Details: Participants were screened for a period up to 28 days prior to Day 1, and then randomized to receive different doses of AMG 404. Cohort 5 was planned but it was never opened.
Groups:
- Cohort 1: Dose Escalation AMG 404 Dose A (Low): Participants received AMG 404 Dose A administered as an IV injection. This cohort contributed to identifying the RP2D.
- Cohort 2: Dose Escalation AMG 404 Dose B (Mid); Cohort 3: Dose Expansion AMG 404 Dose B (Mid): Participants received AMG 404 Dose B administered as an IV injection. This cohort contributed to identifying the RP2D.
- Cohort 4: Dose Exploration AMG 404 Dose C (High): Participants received AMG 404 Dose C administered as an IV injection. This cohort contributed to identifying the RP2D.
- Cohort 6: Dose Expansion AMG 404 RP2D: Participants received AMG 404 at the RP2D (Dose B).
- Cohort 7: AMG 404 RP2D Tumor Specific Efficacy: Participants affected by various types of specific tumors received AMG 404 at the RP2D (Dose B).
- Cohort 8: AMG 404 RP2D Tumor Specific Efficacy: Participants affected by MSI-high and dMMR types of tumors received AMG 404 at the RP2D (Dose B).
- Cohort 9: AMG 404 RP2D Tumor Specific Efficacy: Participants affected by PD-L1 positive non-small cell lung cancer with a TPS ≥ 50% received AMG 404 at the RP2D (Dose B).
Period: Overall Study
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy
Started | 3 | 9 | 21 | 21 | 20 | 42 | 42 | 13
Did Not Receive AMG 404 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Completed | 1 | 4 | 11 | 9 | 14 | 14 | 17 | 3
Not Completed | 2 | 5 | 10 | 12 | 6 | 28 | 25 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 1 | 4 | 5 | 3
Not completed — Decision by Sponsor | 0 | 0 | 1 | 0 | 1 | 1 | 10 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Death | 2 | 5 | 8 | 10 | 3 | 20 | 10 | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who received at least one dose of AMG 404.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy | Total
Number analyzed (Participants) | 3 | 9 | 21 | 21 | 20 | 42 | 42 | 13 | 171
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 59.3 (10.7) | 62.1 (9.8) | 59.3 (14.5) | 58.8 (12.6) | 60.1 (8.7) | 59.5 (14.5) | 62.5 (11.8) | 64.6 (9.0) | 60.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 10 | 11 | 10 | 17 | 23 | 2 | 79
  Male | 2 | 4 | 11 | 10 | 10 | 25 | 19 | 11 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 1 | 0 | 7 | 1 | 13
  Not Hispanic or Latino | 1 | 9 | 20 | 19 | 19 | 37 | 35 | 12 | 152
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 5 | 4 | 4 | 8 | 11 | 9 | 41
  Black (or African American) | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 7
  Multiple | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 9 | 14 | 14 | 15 | 28 | 28 | 3 | 113
  Other | 0 | 0 | 1 | 1 | 1 | 6 | 0 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: Toxicities were graded with the Common Terminology Criteria for Adverse Events CTCAE v5.0., the following toxicities were classified as DLTs:
  * Any treatment related grade 5 toxicity
  * Grade 4 neutropenia or thrombocytopenia
  * Febrile neutropenia
  * Grade 4 anemia
  * Grade 3 or 4 non-hematologic toxicity
  * Recurrent grade 2 pneumonitis
  * Any other toxicity requiring permanent discontinuation of AMG 404.
Time Frame: Up to Day 28
Population: The DLT analysis set included DLT evaluable participants who had completed the DLT window period of 28 days on AMG 404 treatment (starting cycle 1, day 1) or experienced a DLT any time during the DLT window or had received at least 90% of the planned dose of investigational product and was followed for at least 1 cycle. Only participants in cohort 1 to 4 were DLT-evaluable.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High)
Number analyzed (Participants) | 3 | 7 | 4 | 13
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is any adverse event (AE) starting on or after the first administration of investigational product (IP) and up to and including 140 days after the last IP dose date or end of the study, whichever occurs earlier. A TEAE with unknown/missing relatedness to AMG 404 is assumed as an event is related to AMG 404. A serious adverse event (SAE) is defined as an adverse event that: is fatal, is life threatening, requires in-patient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and other medically important serious event. A treatment-related AE (TRAE) is any TEAE that per investigator review has a reasonable possibility of being caused by the investigational product. In the unlikely event that the relationship is missing, the TEAE will be considered TRAE and documented in a footnote of the treatment-related summary.
Time Frame: Up to the last dose of AMG 404 + 140 days (approximately 46 months); median (min, max) exposure to AMG 404 was 3.58 (0.02, 41.7) months
Population: The safety analysis set consisted of all participants who received at least one dose of AMG 404.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy
Number analyzed (Participants) | 3 | 9 | 20 | 21 | 20 | 41 | 41 | 13
Participants
  All TEAEs | 3 | 9 | 20 | 21 | 20 | 41 | 40 | 13
  Fatal AEs | 1 | 4 | 3 | 8 | 2 | 15 | 7 | 5
  SAEs | 2 | 5 | 12 | 15 | 11 | 28 | 16 | 7
  TRAEs | 1 | 5 | 8 | 15 | 13 | 34 | 26 | 8

3. Secondary Outcome: AMG 404 Pharmacokinetic (PK) Parameter by Dose Group: Maximum Observed Serum Concentration (Cmax) During Cycle 1 and 2
Description: Maximum concentration of AMG 404 in blood serum at different time points.
Time Frame: Day 1 pre-dose, end of infusion (EOI), 2h, 4h post dose; Day 2; Day 4; Day 8; Day 15 of Cycle 1 and 2 (28 day cycle length)
Population: The PK Analysis Set contained all participants who received at least 1 dose of AMG 404 and had at least 1 PK sample collected. These participants were evaluated for PK analysis unless the number of data points required for analysis was not enough, or significant protocol deviations affected the data, or if key dosing or sampling information was missing. Per SAP, cohorts have been combined by dose for reporting of PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- AMG 404 Dose A (Low) Q4W: Participants who received AMG 404 Dose A during the treatment period.
- AMG 404 Dose B (Mid) Q4W: Participants who received AMG 404 Dose B during the treatment period.
- AMG 404 Dose C (High) Q4W: Participants who received AMG 404 Dose C during the treatment period.
Arm/Group | AMG 404 Dose A (Low) Q4W | AMG 404 Dose B (Mid) Q4W | AMG 404 Dose C (High) Q4W
Number analyzed (Participants) | 3 | 126 | 21
µg/mL
  Cycle 1 | 84 (38) | 176 (23) | 398 (24)
  Cycle 2: number analyzed (Participants) | 3 | 112 | 16
  Cycle 2 | 96 (39) | 203 (33) | 485 (50)

4. Secondary Outcome: AMG 404 PK Parameter by Dose Group: Time to Achieve Cmax (Tmax) During Cycle 1 and 2
Description: Tmax represents the time to reach Cmax in the blood serum.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: Hour
Arm/Group | AMG 404 Dose A (Low) Q4W | AMG 404 Dose B (Mid) Q4W | AMG 404 Dose C (High) Q4W
Number analyzed (Participants) | 3 | 126 | 21
Hour
  Cycle 1 | 0.550 [0.550 to 0.667] | 0.783 [0.317 to 25.3] | 2.50 [0.533 to 72.6]
  Cycle 2: number analyzed (Participants) | 3 | 112 | 16
  Cycle 2 | 2.53 [0.967 to 2.57] | 0.742 [0.500 to 72.9] | 0.883 [0.500 to 4.75]

5. Secondary Outcome: AMG 404 PK Parameter by Dose Group: Area Under the Serum Concentration-time Curve From Day 0 to Day 28 (AUC0-28d) During Cycle 1 and 2
Description: Assessment of AMG 404 exposure over 28 days.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/mL
Arm/Group | AMG 404 Dose A (Low) Q4W | AMG 404 Dose B (Mid) Q4W | AMG 404 Dose C (High) Q4W
Number analyzed (Participants) | 3 | 126 | 21
day*µg/mL
  Cycle 1: number analyzed (Participants) | 3 | 124 | 20
  Cycle 1 | 732 (40) | 1660 (30) | 3800 (31)
  Cycle 2: number analyzed (Participants) | 3 | 108 | 16
  Cycle 2 | 1130 (27) | 2240 (33) | 4730 (49)

6. Secondary Outcome: Number of Participants With Anti-AMG 404 Antibodies
Description: Transient was defined as the number of participants with negative result at the participant's last time point tested within the study period. Only participants with both baseline and post-baseline are included.
Time Frame: Day 1 pre-dose and Day 15
Population: The safety analysis set consisted of all participants who received at least one dose of AMG 404.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy
Number analyzed (Participants) | 3 | 9 | 20 | 21 | 20 | 41 | 41 | 13
Participants
  Positive at anytime | 0 | 1 | 4 | 1 | 4 | 11 | 7 | 2
  Positive at or before baseline | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Positive post-baseline and negative at baseline: number analyzed (Participants) | 3 | 7 | 20 | 19 | 19 | 41 | 38 | 13
  Positive post-baseline and negative at baseline | 0 | 1 | 3 | 1 | 4 | 11 | 5 | 2
  Transient: number analyzed (Participants) | 3 | 7 | 20 | 19 | 19 | 41 | 38 | 13
  Transient | 0 | 1 | 1 | 0 | 4 | 7 | 4 | 2

7. Secondary Outcome: Objective Tumor Response Per Evaluation Criteria in Solid Tumours (RECIST) V1.1
Description: Objective response was defined as a tumor response assessment of either complete response (CR) (disappearance of all target lesions) or partial response (PR) (at least a 30% decrease in the sum of the diameters of target lesions) measured by positron emission tomography(PET)/computed tomography (CT), CT or magnetic resonance imaging (MRI) and assessed per RECIST v1.1. Participants who did not experience PR/CR or did not have any follow-up tumor assessments was regarded as non-responders. This endpoint was determined only for participants with measurable disease at baseline.
Time Frame: Up to approximately 54 months
Population: The safety analysis set consisted of all participants who received at least one dose of AMG 404.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy
Number analyzed (Participants) | 3 | 9 | 20 | 21 | 20 | 41 | 41 | 13
Percentage of participants | 0.0 [0.00 to 53.58] | 0.0 [0.00 to 22.57] | 5.0 [0.53 to 18.10] | 4.8 [0.50 to 17.29] | 25.0 [12.69 to 41.49] | 17.1 [9.76 to 27.04] | 36.6 [26.44 to 47.78] | 30.8 [14.16 to 52.34]

8. Secondary Outcome: Duration of Response (DOR) Per Modified RECIST v1.1
Description: DOR was defined as the time from the first documentation of objective response (CR or PR) until the first documentation of disease progression or death due to any cause, whichever occurred first. Only participants who achieved objective response were evaluated for DOR. DOR was censored at the last evaluable post-baseline tumor assessment date; otherwise, at the first dose of IP.
  Kaplan-Meier (KM) analysis was used to estimate DOR for responders, providing a median value and 80% confidence intervals (CI) where sufficient data were available. The Brookmeyer and Crowley method was used to calculate confidence intervals. For cohorts with limited responders or heavily censored data, the median DOR or CI bounds could not be calculated.
Time Frame: Up to approximately 43 months
Population: The safety analysis set included all participants who received at least one dose of AMG 404. The DOR analysis was conducted for participants who achieved an objective response (CR or PR) as determined by modified RECIST 1.1 criteria. Participants who did not achieve an objective response were not included in the DOR analysis, as DOR could not be calculated for these cases.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 5 | 7 | 15 | 4
Months |  |  | NA [NA to NA] — Median and CI could not be calculated due to the low number of observations. | 16.85 [NA to NA] — The lower and upper CIs could not be calculated as only one participant had an OR and contributed to the DOR analysis. | NA [5.55 to NA] — Median and upper CI could not be calculated due to the low number of observations. | 11.07 [5.55 to 20.24] | NA [25.76 to NA] — Median and upper CI could not be calculated due to the low number of observations. | NA [2.66 to NA] — Median and upper CI could not be calculated due to the low number of observations.

9. Secondary Outcome: Disease Control Rate (DCR) Per Modified RECIST v1.1
Description: DCR was defined as the percentage of participants in whom objective response (CR or PR) or stable disease (SD) was determined as per RECIST v1.1.
Time Frame: Up to approximately 54 months
Population: The safety analysis set consisted of all participants who received at least one dose of AMG 404.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy
Number analyzed (Participants) | 3 | 9 | 20 | 21 | 20 | 41 | 41 | 13
Percentage of participants | 33.3 [3.45 to 80.42] | 44.4 [21.04 to 69.90] | 35.0 [20.67 to 51.80] | 42.9 [27.78 to 59.05] | 55.0 [38.48 to 70.71] | 48.8 [37.81 to 59.85] | 70.7 [59.76 to 80.07] | 76.9 [55.57 to 91.20]

10. Secondary Outcome: Duration of Stable Disease (DoSD) Per Modified RECIST v1.1
Description: DoSD was measured from the start of treatment until the first documentation of disease progression or death due to any cause. DoSD was calculated only in participants with the best overall response of SD, defined as neither sufficient shrinkage to qualify PR nor sufficient increase to qualify for PD.
  KM analysis was used to estimate the median DoSD, and CIs were calculated using the Brookmeyer and Crowley method. DoSD was censored at the last evaluable post-baseline tumor assessment date or at the first dose of IP, if no progression or death was documented.
Time Frame: Up to approximately 54 months
Population: The analysis population consisted of participants who achieved a best overall response of SD per Modified RECIST v1.1 criteria. This analysis includes only participants from the safety analysis set who received at least one dose of AMG 404 and met the criteria for SD based on tumor assessments.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy
Number analyzed (Participants) | 1 | 4 | 6 | 8 | 6 | 13 | 14 | 6
Months | 5.36 [NA to NA] — The lower and upper confidence intervals could not be calculated because only one participant had a best overall response of SD and contributed to the DoSD analysis. Additionally, there were not enough events at later times to estimate an upper bound. | 5.54 [3.65 to NA] — Upper CI could not be calculated due to the low number of observations. Additionally, there were not enough events at later times to estimate an upper bound. | 6.54 [3.55 to 7.26] | 5.59 [4.11 to NA] — Upper CI could not be calculated due to the low number of observations. Additionally, there were not enough events at later times to estimate an upper bound. | 4.62 [3.61 to 9.46] | 5.55 [4.30 to 5.59] | 16.56 [9.03 to NA] — Upper CI could not be calculated due to the low number of observations. Additionally, there were not enough events at later times to estimate an upper bound. | 3.55 [2.23 to 9.66]

11. Secondary Outcome: Progression-free Survival (PFS) Per Modified RECIST v1.1
Description: PFS was defined as the time from the first dose of IP unite the first documentation of radiological disease progression or death due to any cause, whichever occurred first in the absence of subsequent anticancer therapy.
Time Frame: Up to approximately 48 months
Population: The safety analysis set consisted of all participants who received at least one dose of AMG 404.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy
Number analyzed (Participants) | 3 | 9 | 20 | 21 | 20 | 41 | 41 | 13
Months | 2.89 [1.48 to NA] — Upper CI could not be calculated due to the low number of observations. | 1.84 [1.41 to 3.71] | 1.89 [1.84 to 3.55] | 1.84 [1.68 to 4.50] | 3.68 [2.53 to 9.46] | 3.06 [1.87 to 4.30] | 16.56 [9.03 to 29.24] | 4.37 [2.23 to 14.98]

ADVERSE EVENTS:
Time Frame: Up to approximately 54 months
Description: All-cause mortality was collected for all enrolled participants; AE/SAE was collected for all participants who received at least 1 dose of AMG 404.
Groups:
- Overall Subjects: Overall Subjects
Arm/Group | Cohort 1: Dose Escalation AMG 404 Dose A (Low) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) | Cohort 4: Dose Exploration AMG 404 Dose C (High) | Cohort 6: Dose Expansion AMG 404 RP2D | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy | Overall Subjects
All-Cause Mortality (participants affected / at risk) | 2/3 | 5/9 | 8/21 | 10/21 | 3/20 | 20/42 | 10/42 | 5/13 | 63/171
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/9 | 12/20 | 15/21 | 11/20 | 28/41 | 16/41 | 7/13 | 96/168
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 20/20 | 20/21 | 20/20 | 41/41 | 39/41 | 12/13 | 164/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Dose Escalation AMG 404 Dose A (Low) (N=3) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) (N=9) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) (N=20) | Cohort 4: Dose Exploration AMG 404 Dose C (High) (N=21) | Cohort 6: Dose Expansion AMG 404 RP2D (N=20) | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy (N=41) | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy (N=41) | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy (N=13) | Overall Subjects (N=168)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Addison's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 5
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin graft failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Wound haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Dedifferentiated liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Keratinising squamous cell carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Malignant sweat gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nasopharyngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Testicular germ cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Thymic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Undifferentiated sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 5
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Device occlusion (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Severe cutaneous adverse reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Dose Escalation AMG 404 Dose A (Low) (N=3) | Cohort 2: Dose Escalation AMG 404 Dose B (Mid) (N=9) | Cohort 3: Dose Expansion AMG 404 Dose B (Mid) (N=20) | Cohort 4: Dose Exploration AMG 404 Dose C (High) (N=21) | Cohort 6: Dose Expansion AMG 404 RP2D (N=20) | Cohort 7: AMG 404 RP2D Tumor Specific Efficacy (N=41) | Cohort 8: AMG 404 RP2D Tumor Specific Efficacy (N=41) | Cohort 9: AMG 404 RP2D Tumor Specific Efficacy (N=13) | Overall Subjects (N=168)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 3 | 5 | 7 | 6 | 2 | 29
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 0 | 7
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Addison's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 3 | 0 | 8
Hypothyroidism (Endocrine disorders) | 0 | 1 | 2 | 3 | 2 | 4 | 4 | 0 | 16
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 6
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 5
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 4 | 0 | 9
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 5 | 4 | 3 | 3 | 5 | 0 | 21
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 2 | 0 | 5 | 0 | 11
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 4 | 9 | 9 | 3 | 33
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 6 | 1 | 5 | 4 | 12 | 1 | 31
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 5
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 5
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 5 | 7 | 5 | 7 | 9 | 13 | 1 | 49
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4 | 2 | 2 | 6 | 7 | 4 | 1 | 26
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 7
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 1 | 9
Chills (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 4 | 6 | 7 | 7 | 14 | 18 | 2 | 60
Hernia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 6
Oedema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 1 | 1 | 1 | 1 | 0 | 5 | 2 | 1 | 12
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 6
Pyrexia (General disorders) | 0 | 1 | 4 | 3 | 3 | 8 | 6 | 5 | 30
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Contrast media reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 12 | 3 | 18
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 4
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 4
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 6
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 5
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 2 | 2 | 2 | 7 | 0 | 16
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 1 | 3 | 3 | 6 | 0 | 16
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 4
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 8
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Urethral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 0 | 1 | 2 | 3 | 2 | 11
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 4 | 0 | 1 | 3 | 4 | 2 | 15
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 1 | 3 | 0 | 8
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 4
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 6
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 4
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 1 | 2 | 3 | 1 | 11
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 4 | 8 | 5 | 9 | 8 | 4 | 41
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 3 | 1 | 1 | 0 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 4 | 10 | 10 | 0 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1 | 6 | 10 | 0 | 21
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1 | 3 | 1 | 0 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0 | 6 | 5 | 0 | 15
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 4
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 3 | 7 | 3 | 0 | 15
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 4
Headache (Nervous system disorders) | 0 | 0 | 0 | 3 | 2 | 5 | 5 | 0 | 15
Hemianopia homonymous (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 5
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 5
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 4
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 4 | 0 | 8
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 3 | 0 | 3 | 7 | 2 | 18
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 5
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 0 | 3 | 5 | 1 | 15
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 3 | 9 | 3 | 1 | 20
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 7
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 4
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 7
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 5
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 4 | 1 | 4 | 11 | 2 | 23
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 2 | 8 | 6 | 2 | 23
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 5 | 1 | 9
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 7
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 5
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03853109/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03853109/SAP_001.pdf